CLINICAL TRIAL: NCT00861562
Title: Clinical Efficacy and Safety Evaluation of the Drug Imescard Compound Water Smartweed Pills
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Paulo Dornelles Picon, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04372
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Constipation; Hemorrhoids
Keywords: constipation; hemorrhoids; water smartweed; RCT
MeSH Terms: conditions — Hemorrhoids; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imescard pills/Placebo crossover (Active Comparator): Patients received Imescard water smartweed composed pills during the first intervention period and placebo during the second, after a 10-day washout period.
  Interventions: Drug: Imescard water smartweed composed pills; Drug: Placebo
- Placebo/Imescard pills crossover (Active Comparator): Patients received placebo during the first intervention period and Imescard water smartweed composed pills during the second, after a 10-day washout period.
  Interventions: Drug: Imescard water smartweed composed pills; Drug: Placebo

INTERVENTIONS:
Drug: Imescard water smartweed composed pills — 01 pill at every 8 hours for 5 days.
Drug: Placebo — 01 pill at every 8 hours for 5 days, with the exact same appearance as the other intervention.

SUMMARY:
The purpose of this study was to assess the clinical efficacy and safety of the drug Imescard water smartweed compound pills in the treatment of patients with chronic constipation and hemorrhoidal disease.

DETAILED DESCRIPTION:
The Imescard compound water smartweed pills are currently registered in Brazil at the National Sanitary Surveillance Agency (ANVISA) as a laxative for the treatment of constipation, and as a supporting drug in hemorrhoid treatment. Though water smartweed (Polygonum hydropiperoides) has been used throughout the years as an antiinflammatory and in hemorrhoidal treatment, there are no reliable pharmacologic and clinical evidence that demonstrate its efficacy.

The aim of this study was to assess the clinical efficacy and safety of the drug Imescard compound water smartweed pills in the treatment of chronic constipation and hemorrhoidal disease in a randomized, double-blind, crossover, placebo-controlled clinical trial.

Volunteers underwent a clinical evaluation and laboratory exams at enrollment, and 56 patients met the inclusion criteria and agreed to sign the informed consent form. Participants were then randomized into two groups to receive either Imescard pills or placebo, identical in appearance, once at every 8 hours for five days, followed by a 10-day washout period, and then received the other intervention for another 5-day period.

Followup visits were performed at day 1, 5, 15, and 19. At the beginning of each intervention period(days 1 and 15), patients were given diaries that included two questionnaires for each day of treatment, concerning constipation and hemorrhoidal symptoms, and received the intervention, unaware of its content. Colonic transit time was assessed at the end of each intervention period (days 5 and 19) through standard radiologic technique, and laboratory exams were taken three days later. Clinical evaluation and adverse effects assessment was performed at every visit by blinded investigator, and patients also fulfilled WHOQOL Brief, for life quality assessment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 50;
* chronic constipation diagnosis by the American Association of Gastroentherology (AAG) criteria;
* clinical diagnosis of first and second degree hemorrhoids;
* good understanding and collaboration skills;
* correct fulfilling of the questionnaire at recruiting phase;
* absence of abnormalities in laboratory exams at recruiting phase;
* proper use of anticonceptives, in the case of women in fertile age;
* possibility of abstaining from other drugs (including non-medical ones) other than the intervention during the study, except in case of emergency and with the awareness of the responsible party in the study;
* signing informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* known hypersensitivity to any of the intervention's components;
* use of alcohol or illicit substances;
* clinical evidence of immunosuppression;
* diagnosis of any acute disease in activity or exacerbation of a chronic condition(uncontrolled), such as systemic arterial hypertension, ischemic cardiopathy, angle closure glaucoma, symptomatic prostatic hyperplasia, other concomitant anal disease as fissures, abscesses,fistulas,inflammatory bowel disease or colonic and rectal cancer, as well as any other condition that, in the investigator's opinion, may modify the study results unduly to the intervention being tested or that may put the patient in significant risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in colonic transit time assessed through radiologic technique. | Day 5 and day 19.

SECONDARY OUTCOMES:
Daily evaluation of constipation and hemorrhoidal symptoms assessed by questionnaires. | Daily from day 1 to 5 and from day 15 to 19.
Health quality improvement assessed by WHOQOL Brief at every followup visit. | Days 1, 5, 15 and 19.
Adverse effects assessed by the investigator, blinded to the intervention, at every followup visit, through physical examination and laboratory exams. | Days 1, 5, 15 and 19.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil